CLINICAL TRIAL: NCT05811026
Title: An Open-Label, Single Center Clinical Study to Evaluate the Efficacy of Periorbital Rejuvenation With a 1927 nm Diode Laser Treatment
Brief Title: Efficacy of Periorbital Rejuvenation With a 1927 nm Diode Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: BRIDGECON CO,.LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202207219DSC
Record Dates: First submitted 2023-03-13; First posted 2023-04-13 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-03

CONDITIONS: Laser; Periorbital
Keywords: 1927 nm; periorbital rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm A: 2-week interval between treatments (Experimental): The interval between the first, second, and third treatments in this arm is two weeks, and the follow-up session will take place four weeks after the third treatment.
  Interventions: Device: Periorbital rejuvenation with a 1927 nm diode laser treatment (2-week interval)
- Arm B: 4-week interval between treatments (Experimental): The interval between the first, second, and third treatments in this arm is four weeks, and the follow-up session will take place four weeks after the third treatment.
  Interventions: Device: Periorbital rejuvenation with a 1927 nm diode laser treatment (4-week interval)

INTERVENTIONS:
Device: Periorbital rejuvenation with a 1927 nm diode laser treatment (2-week interval) — * Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W2): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W8): Four weeks after the third treatment, a follow-up assessment will be performed
  Arms: Arm A: 2-week interval between treatments
Device: Periorbital rejuvenation with a 1927 nm diode laser treatment (4-week interval) — * Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W8): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W12): Four weeks after the third treatment, a follow-up assessment will be performed
  Arms: Arm B: 4-week interval between treatments

SUMMARY:
The purpose of this research project is to investigate the treatment design, therapeutic effects and safety of the 1927 nm laser for the rejuvenation of the skin around the eyes.

DETAILED DESCRIPTION:
The chromophore of the 1927 nm diode laser is mainly water, which can be used for skin rejuvenation. This study intends to use the Solta CLEAR+BRILLIANT Laser System, featuring a 1927 nm diode laser with 5 mJ energy, a treatment spot of 140 μm, a treatment depth of 170 μm, and a treatment coverage of approximately 5% per energy level after four rounds of treatment using the patented Intelligent Optical Tracking® System (IOTs). The purpose of this research project is to investigate the treatment design, therapeutic effects and safety of the 1927 nm laser for the rejuvenation of the skin around the eyes. This is an open-label, single-center clinical trial. Participants will be randomized into treatment groups, including Group A (treatment interval of 2 weeks) or Group B (treatment interval of 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. aged between 30 and 65 years old;
2. no significant skin lesions or inflammation on the facial skin;
3. willing and able to comply with study requirements, instructions, and restrictions;
4. signed informed consent form.

Exclusion Criteria:

1. underwent facial active treatment, such as using laser, intense pulsed light, radiofrequency skin tightening, ultrasound skin tightening, botulinum toxin, or dermal fillers injection, within the previous six months;
2. have chronic skin diseases such as atopic dermatitis, psoriasis, chronic urticaria, vitiligo, rosacea, or keloid;
3. pregnant or breastfeeding;
4. suffered from acute illnesses or infections requiring treatment within 14 days before entering the study;
5. have had serious illnesses (such as heart disease, lung disease, brain disease, or liver disease) within the previous three months;
6. allergic to Lidocaine or Prilocaine used in topical anesthetic cream or suffer from methemoglobinemia;
7. used any skin medication on the face within 30 days before the trial, deemed by the principal investigator to affect the study results;
8. deemed unsuitable for the study by the principal investigator.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, MD/PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: 2-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is two weeks, and the follow-up session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (2-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W2): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W8): Four weeks after the third treatment, an end-of-study assessment will be performed
- Arm B: 4-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is four weeks, and the follow-up session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (4-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W8): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W12): Four weeks after the third treatment, an end-of-study assessment will be performed
Period: Overall Study
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [48 to 56.75] | 45 [44.25 to 47.5] | 48 [45 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Texture Score at Visit 4 (End-of-study Session)
Description: The texture score is a parameter measured by the Antera 3D system, calculated based on average roughness (Ra [μm]). Ra roughness, or average roughness, is a standard metric used to describe surface smoothness. It represents the average height of microscopic peaks and valleys on the skin surface. The Ra [μm] values range from 0 to infinity.
  To interpret the texture score, skin surface roughness is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer skin texture. The overall texture score ranges from 0 to infinity.
  Change from baseline in texture score at Visit 4 = texture score at Visit 4 - texture score at baseline
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 0.25 [-0.375 to 7.125] | -4.75 [-7.25 to -0.5]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.075, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 5 — Differece = (2-week interval group) - (4-week interval group)

2. Secondary Outcome: Change From Baseline in Color Measurements (L*) at Visit 4 (End-of-study Session)
Description: In the CIELAB color space, the L* value represents the lightness of a color, indicating how light or dark it appears. The scale ranges from 0 (black) to 100 (white), providing a standardized measure of brightness that aligns with human visual perception. This metric is particularly useful in assessing skin tone. The average L* value within a region of interest was calculated at each visit.
  Change from baseline in L* at Visit 4 = L* at Visit 4 - L* at baseline
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Arm A: 2-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is two weeks, and the follow-up session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (2-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W2): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W8): Four weeks after the third treatment, a follow-up assessment will be performed
- Arm B: 4-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is four weeks, and the follow-up session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (4-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W8): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W12): Four weeks after the third treatment, a follow-up assessment will be performed
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | -0.61495 [-1.0353375 to -0.119875] | -0.798575 [-0.9895125 to -0.1737125]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.4727, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 0.17 — Differece = (2-week interval group) - (4-week interval group)

3. Secondary Outcome: Change From Baseline in Pigmentation Score at Visit 4 (End-of-study Session)
Description: The pigmentation score is a parameter measured by the Antera 3D system, calculated based on the variation (arbitrary units) and average level (arbitrary units). Variation (arbitrary units) indicates mean value within the region of interest of all deviations from the pigmentation average level in absolute value. Average level (arbitrary units) indicates the average concentration of pigmentation in the region of interest. To interpret the pigmentation score, skin pigmentation is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer pigmentation conditions. The overall pigmentation score ranges from 0 to infinity.
  Change from baseline in pigmentation score at Visit 4 = pigmentation score at Visit 4 - pigmentation score at baseline
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | -9 [-9.5 to -7] | -7.5 [-10.375 to -4.75]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.7326, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = -1.5 — Differece = (2-week interval group) - (4-week interval group)

4. Secondary Outcome: Change From Baseline in Pores' Index at Visit 4 (End-of-study Session)
Description: The pores' index is an overall score representing skin porosity within the selected region of interest. It incorporates pore depth, size, and density-condensed into a single parameter. This index is particularly useful for the global evaluation of porosity reduction in before-and-after comparisons.
  Formula: Index = (V / S) × 1000 V = total volume of pores in the selected area (mm³) S = selected area (mm²)
  Change from baseline in pores' index at Visit 4 = pores' index at Visit 4-pores' indexe at baseline
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | -0.02675 [-0.1378625 to 0.2650375] | -0.63555 [-0.8427125 to -0.1460625]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0757, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 0.61 — Differece = (2-week interval group) - (4-week interval group)

5. Secondary Outcome: Change From Baseline in Wrinkles' Score at Visit 4 (End-of-study Session)
Description: The wrinkle score is a parameter measured by the Antera 3D system, calculated based on the indentation index (μm). The indentation index (μm) represents the average depth of all points or dents below the surface level. The indentation index (μm) values range from 0 to infinity.
  To interpret the wrinkle score, skin damage is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate more severe wrinkle conditions. The overall wrinkle score ranges from 0 to infinity.
  Change from baseline in wrinkles' score at Visit 4 = wrinkles' score at Visit 4 - wrinkles' score at baseline
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 13 [-0.5 to 39] | -29.75 [-48.75 to -11.375]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0376, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 37.75 — Differece = (2-week interval group) - (4-week interval group)

6. Secondary Outcome: Change From Baseline in Physician Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 4 (End-of-study Session)
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Physician Assessment of GAIS refers to the GAIS score evaluated by the physician.
  Change from Baseline in Physician Assessment of GAIS at Visit 4 is defined as the GAIS score assessed at Visit 4 in comparison to baseline.
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 2.8 [2.4 to 3.0] | 3.0 [2.7 to 3.3]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.3123, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = -0.17 — Differece = (2-week interval group) - (4-week interval group)

7. Secondary Outcome: Change From Baseline in Patient Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 4 (End-of-study Session)
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Patient Assessment of GAIS refers to the GAIS score evaluated by the patient. Change from Baseline in Patient Assessment of GAIS at Visit 4 is defined as the GAIS score assessed at Visit 4 in comparison to baseline.
Time Frame: Group A: baseline and week 8; Group B: baseline and week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 3.0 [2.0 to 3.0] | 2.0 [2.0 to 2.0]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.1009, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = 1 — Differece = (2-week interval group) - (4-week interval group)

8. Secondary Outcome: Change From Baseline in Texture Score at Visit 2
Description: The texture score is a parameter measured by the Antera 3D system, calculated based on average roughness (Ra [μm]). Ra roughness, or average roughness, is a standard metric used to describe surface smoothness. It represents the average height of microscopic peaks and valleys on the skin surface. The Ra [μm] values range from 0 to infinity.
  To interpret the texture score, skin surface roughness is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer skin texture. The overall texture score ranges from 0 to infinity.
  Change from baseline in texture score at Visit 2 = texture score at Visit 2 - texture score at baseline
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 1.5 [-1 to 5.375] | -4 [-8 to -1.625]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0088, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Mean Difference (Net) = 5.5 — Differece = (2-week interval group) - (4-week interval group)

9. Secondary Outcome: Change From Baseline in Color Measurements (L*) at Visit 2
Description: In the CIELAB color space, the L* value represents the lightness of a color, indicating how light or dark it appears. The scale ranges from 0 (black) to 100 (white), providing a standardized measure of brightness that aligns with human visual perception. This metric is particularly useful in assessing skin tone. The average L* value within a region of interest was calculated at each visit.
  Change from baseline in L* at Visit 2 = L* at Visit 2 - L* at baseline
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | -0.4711 [-0.6366375 to -0.0799375] | -0.44215 [-0.5409375 to 0.5504]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.4274, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = -0.03 — Differece = (2-week interval group) - (4-week interval group)

10. Secondary Outcome: Change From Baseline in Pigmentation Score at Visit 2
Description: The pigmentation score is a parameter measured by the Antera 3D system, calculated based on the variation (arbitrary units) and average level (arbitrary units). Variation (arbitrary units) indicates mean value within the region of interest of all deviations from the pigmentation average level in absolute value. Average level (arbitrary units) indicates the average concentration of pigmentation in the region of interest. To interpret the pigmentation score, skin pigmentation is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer pigmentation conditions. The overall pigmentation score ranges from 0 to infinity.
  Change from baseline in pigmentation score at Visit 2 = pigmentation score at Visit 2 - pigmentation score at baseline
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | -0.5 [-1.875 to 0.75] | -2.25 [-5.25 to 1.5]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.6497, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Mean Difference (Net) = 1.75 — Differece = (2-week interval group) - (4-week interval group)

11. Secondary Outcome: Change From Baseline in Pores' Index at Visit 2
Description: The pores' index is an overall score representing skin porosity within the selected region of interest. It incorporates pore depth, size, and density-condensed into a single parameter. This index is particularly useful for the global evaluation of porosity reduction in before-and-after comparisons.
  Formula: Index = (V / S) × 1000 V = total volume of pores in the selected area (mm³) S = selected area (mm²)
  Change from baseline in pores' index at Visit 2 = pores' index at Visit 2 - pores' index at baseline
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 0.126725 [-0.169925 to 0.777575] | -0.4088 [-0.6626875 to -0.3374875]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0006, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 0.54 — Differece = (2-week interval group) - (4-week interval group)

12. Secondary Outcome: Change From Baseline in Wrinkles' Score at Visit 2
Description: The wrinkle score is a parameter measured by the Antera 3D system, calculated based on the indentation index (μm). The indentation index (μm) represents the average depth of all points or dents below the surface level. The indentation index (μm) values range from 0 to infinity.
  To interpret the wrinkle score, skin damage is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate more severe wrinkle conditions. The overall wrinkle score ranges from 0 to infinity.
  Change from baseline in wrinkles' score at Visit 2 = wrinkles' score at Visit 2 - wrinkles' score at baseline
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 11 [1.625 to 40.25] | -23.5 [-43.125 to -17]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0002, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 34.5 — Differece = (2-week interval group) - (4-week interval group)

13. Secondary Outcome: Change From Baseline in Physician Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 2
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Physician Assessment of GAIS refers to the GAIS score evaluated by the physician.
  Change from Baseline in Physician Assessment of GAIS at Visit 2 is defined as the GAIS score assessed at Visit 2 in comparison to baseline.
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 4.0 [3.8 to 4.0] | 4.0 [3.7 to 4.0]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.6231, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = 0 — Differece = (2-week interval group) - (4-week interval group)

14. Secondary Outcome: Change From Baseline in Patient Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 2
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Patient Assessment of GAIS refers to the GAIS score evaluated by the patient. Change from Baseline in Patient Assessment of GAIS at Visit 2 is defined as the GAIS score assessed at Visit 2 in comparison to baseline.
Time Frame: Group A: baseline and week 2; Group B: baseline and week 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 3.0]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.3327, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = 0 — Differece = (2-week interval group) - (4-week interval group)

15. Secondary Outcome: Change From Baseline in Texture Score at Visit 3
Description: The texture score is a parameter measured by the Antera 3D system, calculated based on average roughness (Ra [μm]). Ra roughness, or average roughness, is a standard metric used to describe surface smoothness. It represents the average height of microscopic peaks and valleys on the skin surface. The Ra [μm] values range from 0 to infinity.
  To interpret the texture score, skin surface roughness is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer skin texture. The overall texture score ranges from 0 to infinity.
  Change from baseline in texture score at Visit 3 = texture score at Visit 3 - texture score at baseline
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 2.75 [-3.75 to 4.25] | -4.5 [-8.5 to -3]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0752, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 7.25 — Differece = (2-week interval group) - (4-week interval group)

16. Secondary Outcome: Change From Baseline in Color Measurements (L*) at Visit 3
Description: In the CIELAB color space, the L* value represents the lightness of a color, indicating how light or dark it appears. The scale ranges from 0 (black) to 100 (white), providing a standardized measure of brightness that aligns with human visual perception. This metric is particularly useful in assessing skin tone. The average L* value within a region of interest was calculated at each visit.
  Change from baseline in L* at Visit 3 = L* at Visit 3 - L* at baseline
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 5
score on a scale | -1.1979 [-1.744225 to -0.7522625] | -0.26345 [-0.64905 to 0.0077]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0982, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = -0.94 — Differece = (2-week interval group) - (4-week interval group)

17. Secondary Outcome: Change From Baseline in Pigmentation Score at Visit 3
Description: The pigmentation score is a parameter measured by the Antera 3D system, calculated based on the variation (arbitrary units) and average level (arbitrary units). Variation (arbitrary units) indicates mean value within the region of interest of all deviations from the pigmentation average level in absolute value. Average level (arbitrary units) indicates the average concentration of pigmentation in the region of interest. To interpret the pigmentation score, skin pigmentation is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate poorer pigmentation conditions. The overall pigmentation score ranges from 0 to infinity.
  Change from baseline in pigmentation score at Visit 3 = pigmentation score at Visit 3 - pigmentation score at baseline
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 5
score on a scale | -3 [-5.875 to -0.75] | -2.5 [-5 to 0]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.8541, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = -0.5 — Differece = (2-week interval group) - (4-week interval group)

18. Secondary Outcome: Change From Baseline in Pores' Index at Visit 3
Description: The pores' index is an overall score representing skin porosity within the selected region of interest. It incorporates pore depth, size, and density-condensed into a single parameter. This index is particularly useful for the global evaluation of porosity reduction in before-and-after comparisons.
  Formula: Index = (V / S) × 1000 V = total volume of pores in the selected area (mm³) S = selected area (mm²)
  Change from baseline in pores' index at Visit 3 = pores' index at Visit 3 - pores' index at baseline
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 5
score on a scale | 0.299125 [-0.123325 to 0.41035] | -0.33025 [-0.73005 to -0.1437]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0758, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 0.63 — Differece = (2-week interval group) - (4-week interval group)

19. Secondary Outcome: Change From Baseline in Wrinkles' Score at Visit 3
Description: The wrinkle score is a parameter measured by the Antera 3D system, calculated based on the indentation index (μm). The indentation index (μm) represents the average depth of all points or dents below the surface level. The indentation index (μm) values range from 0 to infinity.
  To interpret the wrinkle score, skin damage is categorized into five intervals: Mild: 0-25, Moderate: 25-50, Advanced: 50-75, Severe: 75-100, Very Severe: >100. Higher scores indicate more severe wrinkle conditions. The overall wrinkle score ranges from 0 to infinity.
  Change from baseline in wrinkles' score at Visit 3 = wrinkles' score at Visit 3 - wrinkles' score at baseline
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 5
score on a scale | 20.25 [-2.5 to 27] | -21.5 [-36.5 to -21]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.066, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Net) = 41.75 — Differece = (2-week interval group) - (4-week interval group)

20. Secondary Outcome: Change From Baseline in Physician Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 3
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Physician Assessment of GAIS refers to the GAIS score evaluated by the physician.
  Change from Baseline in Physician Assessment of GAIS at Visit 3 is defined as the GAIS score assessed at Visit 3 in comparison to baseline.
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 3.5 [3.3 to 3.7] | 3.7 [3.3 to 3.9]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments; Test type: Superiority; p = 0.6961, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = -0.17 — Differece = (2-week interval group) - (4-week interval group)

21. Secondary Outcome: Change From Baseline in Patient Assessment of Global Aesthetic Improvement Score (GAIS), at Visit 3
Description: Global Aesthetic Improvement Score (GAIS) is a standardized 5-point scale used to assess overall aesthetic improvement following a cosmetic treatment. It ranges as follows: 5 - Very Much Improved, 4 - Much Improved, 3 - Improved, 2 - No Change, 1 - Worse Patient Assessment of GAIS refers to the GAIS score evaluated by the patient. Change from Baseline in Patient Assessment of GAIS at Visit 3 is defined as the GAIS score assessed at Visit 3 in comparison to baseline.
Time Frame: Group A: baseline and week 4; Group B: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 3.0 [3.0 to 3.0] | 2.0 [2.0 to 2.0]
Statistical Analysis 1: Comparison: Arm A: 2-week Interval Between Treatments vs Arm B: 4-week Interval Between Treatments; Test type: Superiority; p = 0.0067, Wilcoxon (Mann-Whitney) — Statistical significance was defined as a p-value < 0.05; Median Difference (Final Values) = 1 — Differece = (2-week interval group) - (4-week interval group)

22. Secondary Outcome: Visual Analogue Scale (VAS) During Treatment
Description: The visual analogue scale (VAS) is a psychometric response scale that can be used in questionnaires, which a higher score suggests greater pain intensity. It ranges from 0 to 10 in increments of 1. A score of 0 cm indicates "no pain" and 10 indicates "worst pain imaginable".
Time Frame: Group A: week 0; Group B: week 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
Number analyzed (Participants) | 10 | 10
score on a scale | 5 [4 to 7] | 6.5 [3.5 to 7]

ADVERSE EVENTS:
Time Frame: Arm A: 8 weeks, Arm B: 12 weeks
Groups:
- Arm A: 2-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is two weeks, and the end-of-study session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (2-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W2): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W8): Four weeks after the third treatment, an end-of-study assessment will be performed
  There are a total 30 person-times of treatment.
- Arm B: 4-week Interval Between Treatments: The interval between the first, second, and third treatments in this arm is four weeks, and the end-of-study session will take place four weeks after the third treatment.
  Periorbital rejuvenation with a 1927 nm diode laser treatment (4-week interval): - Visit 1 (W0): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 2 (W4): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 3 (W8): Clear + Brilliant™ Permea device periorbital treatment
  * Visit 4 (W12): Four weeks after the third treatment, an end-of-study assessment will be performed
  There are a total 30 person-times of treatment.
Arm/Group | Arm A: 2-week Interval Between Treatments | Arm B: 4-week Interval Between Treatments
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 2-week Interval Between Treatments (N=10) | Arm B: 4-week Interval Between Treatments (N=10)
Severe erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Severe swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Severe itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Severe tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Severe scaling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05811026/Prot_SAP_001.pdf